CLINICAL TRIAL: NCT00181233
Title: Functional Energetics and Imaging for Phenotypic Characterization of Patients at Risk for Sudden Cardiac Death
Brief Title: Imaging Techniques for Identifying Factors of Sudden Cardiac Death Risk
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Donald W. Reynolds Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00037404
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Sudden Cardiac Death
MeSH Terms: conditions — Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Sudden cardiac death is a tragic event that strikes all age groups and is unfortunately increasing in prevalence. Because it is difficult to predict those at highest risk, this study is designed to test the hypothesis that new imaging techniques (magnetic resonance imaging [MRI] and computed tomography [CT]) are useful for identifying factors which put people at high risk for sudden death.

DETAILED DESCRIPTION:
Some people with heart disease and a weak heart muscle experience abnormal electrical activity of the heart that may predispose them to sudden death. In light of this risk, it has been recommended that such patients undergo implantation of an implantable cardioverter defibrillator (ICD). Your doctors have determined that you are such a patient and are to undergo implantation of an ICD. It is unclear who among the many patients who undergo ICD implantation for this reason are at greatest risk of sudden death and therefore require electrical response from their ICD. This research is being done to determine whether new imaging tests, such as magnetic resonance imaging (MRI) or multi-detector computed tomography (MDCT), can be used to predict who is at highest risk of sudden death and require electrical response from their ICD.

ELIGIBILITY:
Inclusion Criteria:

* Left ventricular ejection fraction <or = 35%
* Planned implantable cardioverter-defibrillator (ICD) implantation for clinical indications (primary prevention)

Exclusion Criteria:

* History of sudden death (secondary prevention)
* Contraindication to undergoing MRI (metallic implant, pacemaker, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with contractile dysfunction (EF< or = 35%) on an ischemic or non-ischemic basis undergoing clinically-indicated ICD implantation for primary prevention of sudden cardiac death (SCD)
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2003-10; Primary Completion 2028-02 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
sudden cardiac death | 6 month intervals
cardiovascular death | 6 month intervals
appropriate ICD discharge | 6 month intervals
composite sudden cardiac death and appropriate ICD discharge | 6 month intervals

SECONDARY OUTCOMES:
heart failure admission | 6 month intervals

OTHER OUTCOMES:
cardiac transplantation | 6 month intervals
myocardial revascularization | 6 month intervals
left ventricular assist device placement | 6 month intervals
biventricular pacemaker placement | 6 month intervals

CONTACTS AND LOCATIONS:
Overall Officials: Katherine C Wu, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Samuel TJ, Lai S, Schar M, Wu KC, Steinberg AM, Wei AC, Anderson ME, Tomaselli GF, Gerstenblith G, Bottomley PA, Weiss RG. Myocardial ATP depletion detected noninvasively predicts sudden cardiac death risk in patients with heart failure. JCI Insight. 2022 Jun 22;7(12):e157557. doi: 10.1172/jci.insight.157557. PMID 35579938
- [Derived] Wu KC, Gerstenblith G, Guallar E, Marine JE, Dalal D, Cheng A, Marban E, Lima JA, Tomaselli GF, Weiss RG. Combined cardiac magnetic resonance imaging and C-reactive protein levels identify a cohort at low risk for defibrillator firings and death. Circ Cardiovasc Imaging. 2012 Mar;5(2):178-86. doi: 10.1161/CIRCIMAGING.111.968024. Epub 2012 Jan 20. PMID 22267750
- [Derived] Wu KC, Weiss RG, Thiemann DR, Kitagawa K, Schmidt A, Dalal D, Lai S, Bluemke DA, Gerstenblith G, Marban E, Tomaselli GF, Lima JA. Late gadolinium enhancement by cardiovascular magnetic resonance heralds an adverse prognosis in nonischemic cardiomyopathy. J Am Coll Cardiol. 2008 Jun 24;51(25):2414-21. doi: 10.1016/j.jacc.2008.03.018. PMID 18565399